CLINICAL TRIAL: NCT07317531
Title: Effects of Expiratory Muscle Training Added to Pulmonary Rehabilitation on Pulmonary Function, Respiratory Muscle Strength, and Functional Capacity in Patients With Bronchiectasis
Brief Title: Effects of Expiratory Muscle Training Added to Pulmonary Rehabilitation in Patients With Bronchiectasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Collaborators: Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Reyhan Kaygusuz, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: bronchiectasis and EMT
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis Adult; Expiratory Muscle Training; Pulmonary Rehabilitation; Lung Function Tests; Functional Capacity; Respiratory Muscle Strength

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, randomized controlled, parallel-group clinical trial. Eligible patients with bronchiectasis will be randomly assigned to either a pulmonary rehabilitation program alone (control group) or pulmonary rehabilitation combined with expiratory muscle training (intervention group). Both groups will receive the same standard pulmonary rehabilitation protocol, while the intervention group will additionally perform structured expiratory muscle training. Outcomes will be assessed at baseline and after completion of the intervention period to compare the effects of the two treatment approaches.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulmonary rehabilitation (Experimental): Participants will receive a standard pulmonary rehabilitation program consisting of aerobic exercise, resistance training, breathing exercises, and patient education.
  Interventions: Other: pulmonary rehabilitation
- Pulmonary Rehabilitation plus Expiratory Muscle Training (Experimental): Participants will receive a standard pulmonary rehabilitation program combined with structured expiratory muscle training.
  Interventions: Other: pulmonary rehabilitation; Device: Expiratory muscle training

INTERVENTIONS:
Other: pulmonary rehabilitation — Participants will undergo a standard pulmonary rehabilitation program including supervised aerobic exercise, resistance training, breathing exercises, and patient education. The program will be conducted three times per week over the intervention period in accordance with current pulmonary rehabilitation guidelines.
Device: Expiratory muscle training — Expiratory muscle training will be performed using an adjustable PowerBreathe EX1 expiratory muscle training device. The initial training load will be set at 30-40% of the participant's maximal expiratory pressure (MEP) and will be progressively increased by 5-10% on a weekly basis. Training sessions will be conducted three days per week, consisting of two sets per day, with each set including 10-15 repetitions.
  Arms: Pulmonary Rehabilitation plus Expiratory Muscle Training

SUMMARY:
This randomized, single-blind, parallel-group controlled trial aims to investigate the effects of expiratory muscle training added to standard pulmonary rehabilitation on respiratory muscle strength, pulmonary function, cough effectiveness, exercise capacity, dyspnea perception, and quality of life in patients with non-cystic fibrosis bronchiectasis. Eligible patients aged 18-70 years with stable disease will be randomly assigned to either a pulmonary rehabilitation-only group or a pulmonary rehabilitation combined with expiratory muscle training group. Outcomes will be assessed at baseline and after completion of the intervention period.

DETAILED DESCRIPTION:
his study will be conducted as a randomized controlled, single-blind, parallel-group trial. Ethical approval has been applied for from the University of Health Sciences Hamidiye Non-Drug and Non-Medical Device Interventional Research Ethics Committee, and the evaluation process is currently ongoing. Upon receipt of the ethical approval, the approval document will be submitted to the Scientific Research Projects (BAP) Commission by the principal investigator.

Following ethical approval, individuals aged 18-70 years with a clinical diagnosis of stable non-cystic fibrosis bronchiectasis who are being followed at the Pulmonary Rehabilitation Unit of the University of Health Sciences Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital will be eligible for inclusion. Patients who have experienced an acute exacerbation within the last three months, have severe cardiac, neurological, or orthopedic diseases, demonstrate lack of cooperation, or have communication difficulties will be excluded from the study.

Eligible participants will be randomly assigned to one of two groups using a simple randomization method: (1) a control group receiving a standard pulmonary rehabilitation program, and (2) an intervention group receiving standard pulmonary rehabilitation combined with expiratory muscle training.

The standard pulmonary rehabilitation program will be conducted on an outpatient basis for eight weeks, three days per week, under direct supervision. Prior to enrollment, all participants will undergo cardiology consultation, lower extremity venous Doppler ultrasonography for deep vein thrombosis screening, chest radiography, electrocardiography, pulmonary function testing, and routine laboratory assessments. Baseline evaluations will include symptom assessment, physical examination, oxygen saturation levels, current medical treatments, comorbidities, disease duration, oxygen therapy requirements, use of respiratory support devices, smoking history, and anthropometric measurements (height, weight, body mass index, and fat-free mass). Pulmonary function tests (FVC, FEV₁, and diffusion capacity), nutritional assessment, medication review and education, disease-related patient and caregiver education, and functional exercise capacity assessment using field tests such as the 6-minute walk test will be performed. All assessments will be repeated at the end of the rehabilitation program. Written informed consent will be obtained from all participants prior to inclusion.

During the eight-week rehabilitation period, participants will attend supervised sessions at the hospital three days per week and will be encouraged to continue prescribed exercises at home on non-supervised days using an exercise diary. Oxygen saturation and heart rate will be continuously monitored using pulse oximetry during sessions, and blood pressure measurements will be taken before and after exercise. Perceived dyspnea and fatigue levels will be assessed using the Borg scale.

Exercise training will be individualized based on baseline exercise capacity assessments. Each session will include upper and lower extremity strengthening exercises, stretching, relaxation exercises, aerobic training (treadmill walking and cycling), breathing exercises, and relaxation techniques. Aerobic exercise will be performed at 60-80% of the target heart rate, consisting of a 10-minute warm-up, 30 minutes of aerobic exercise, and a 10-minute cool-down period. Resistance training will be performed at 50% of one-repetition maximum, with one set of 10 repetitions per session, targeting both upper and lower extremity muscle groups.

In addition to pulmonary rehabilitation, participants in the intervention group will perform expiratory muscle training using an adjustable PowerBreathe EX1 expiratory muscle training device. The initial training resistance will be set at 30-40% of maximal expiratory pressure (MEP) and will be progressively increased by 5-10% on a weekly basis. Training will be performed three days per week, consisting of two sets per day, with each set including 10-15 repetitions.

Outcome measures will be assessed at baseline and after completion of the intervention period by an experienced physiotherapist using standardized procedures in accordance with international guidelines. Pulmonary function will be assessed using spirometry to measure forced vital capacity (FVC), forced expiratory volume in one second (FEV₁), and the FEV₁/FVC ratio, following American Thoracic Society (ATS) and European Respiratory Society (ERS) standards. Peak cough flow will be measured in liters per minute using a peak flow meter. Respiratory muscle strength will be evaluated by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using a digital manometer in accordance with ATS/ERS guidelines. Functional exercise capacity will be assessed using the 6-minute walk test performed on a 30-meter corridor according to ATS protocol, with continuous monitoring of oxygen saturation, heart rate, and perceived exertion using the Borg scale. Dyspnea severity will be evaluated using the modified Medical Research Council (mMRC) dyspnea scale. Health-related quality of life will be assessed using the St. George's Respiratory Questionnaire (SGRQ). Fatigue severity will be evaluated using the Fatigue Severity Scale.

Statistical analysis will be performed using SPSS software. Normally distributed data will be analyzed using independent and paired t-tests, while non-normally distributed data will be analyzed using the Mann-Whitney U test and Wilcoxon signed-rank test. Statistical significance will be set at p < 0.05. Sample size was determined using power analysis with G*Power version 3.1.9.7. Based on an effect size of 0.25, a significance level of 0.05, and a power of 0.80, a total sample size of 34 participants was calculated. Considering a potential dropout rate of 15%, the total sample size was increased to 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years

  * Clinical diagnosis of non-cystic fibrosis bronchiectasis
  * Stable disease status
  * Follow-up at the Pulmonary Rehabilitation Unit of University of Health Sciences Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital
  * Ability to understand and comply with the study procedures
  * Provided written informed consent

Exclusion Criteria:

* Acute exacerbation within the last 3 months
* Diagnosis of cystic fibrosis-related bronchiectasis
* Presence of severe cardiac, neurological, or orthopedic diseases that may interfere with exercise training
* Cognitive impairment, lack of cooperation, or communication difficulties
* Any medical condition contraindicating participation in pulmonary rehabilitation or expiratory muscle training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Baseline and 8 weeks
  Functional capacity will be evaluated using the 6-minute walk test (6MWT) performed on a 30-meter corridor in accordance with ATS guidelines. Total walking distance will be recorded as the primary outcome of the test.
Maximum Inspiratory Pressure (MIP) | Baseline and 8 weeks
  Respiratory muscle strength will be assessed using maximum inspiratory pressure (MIP), measured with a portable mouth pressure device according to standard guidelines. Higher values indicate better inspiratory muscle function.
Maximum Expiratory Pressure (MEP) | Baseline and 8 weeks
  Respiratory muscle strength will be assessed using maximum expiratory pressure (MEP), measured with a portable mouth pressure device according to standard guidelines. Higher values indicate better expiratory muscle function.
Forced Vital Capacity (FVC) | Baseline and 8 weeks
  Forced Vital Capacity (FVC) will be measured using a portable spirometer calibrated according to American Thoracic Society (ATS) and European Respiratory Society (ERS) standards. The best result from at least three attempts will be recorded.
Forced Expiratory Volume in 1 Second (FEV₁) | Baseline and 8 weeks
  Forced Expiratory Volume in 1 second (FEV₁) will be measured using a portable spirometer calibrated according to ATS/ERS standards. The best result from at least three attempts will be recorded.
FEV₁/FVC Ratio | Baseline and 8 weeks
  FEV₁/FVC ratio will be calculated from spirometry results. The best result from at least three attempts will be recorded.
Cough Strength (Peak Cough Flow, PCF) | Baseline and 8 weeks
  Peak Cough Flow (PCF) will be measured using a peak flow meter.

SECONDARY OUTCOMES:
Dyspnea Severity | Baseline and 8 weeks
  Dyspnea severity will be evaluated using the modified Medical Research Council (mMRC) dyspnea scale, ranging from 0 (no dyspnea) to 4 (severe dyspnea).
Health-Related Quality of Life | Baseline and 8 weeks
  Quality of life will be evaluated using the St. George's Respiratory Questionnaire (SGRQ), including symptom, activity, and impact domains. Higher scores indicate worse health status.Scores for each domain and the total score range from 0 to 100, with higher scores indicating poorer health-related quality of life.
Fatigue Severity | Baseline and 8 weeks
  Fatigue severity will be assessed using the Fatigue Severity Scale (FSS), a validated self-report questionnaire evaluating the impact of fatigue on daily functioning.The scale consists of nine items scored from 1 to 7, with higher scores indicating greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: reyhan kaygusuz benli, Asst Prof, Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided